CLINICAL TRIAL: NCT01289925
Title: Antioxidant Nutrient Inflammation Interventions in Older Adults
Brief Title: Effect of Selenium Intervention on Inflammation in Older Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NA_00002109
Record Dates: First submitted 2011-02-03; First posted 2011-02-04 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Inflammation
Keywords: dietary supplement; selenium; healthy volunteer; Johns Hopkins; older; aging; geriatrics; baltimore; mineral; over 70
MeSH Terms: conditions — Inflammation; Calcinosis | interventions — Selenium; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Selenium (Experimental)
  Interventions: Dietary Supplement: Selenium
- Sugar Pill (Placebo Comparator)
  Interventions: Other: Sugar Pill Placebo

INTERVENTIONS:
Dietary Supplement: Selenium — 200 micrograms of selenium (in the form of selenium methionine) in tablet form taken orally daily for 8 weeks. Capsule molds with inert coating.
  Arms: Selenium
Other: Sugar Pill Placebo — Placebo supplements in the same capsule mold as selenium and coated with the same inert coating. 1 tablet daily for 8 weeks.
  Arms: Sugar Pill

SUMMARY:
Serum levels of inflammatory mediators increase with age and are strongly associated with the most common and the most devastating health conditions found in older adults including frailty, chronic disease, disability and increased mortality. Even though the processes that contribute to increased inflammatory mediators are likely not completely reversible in older adults, the development of a safe and effective intervention that modulates inappropriate inflammatory responses could be a very important component of prevention against frailty and other adverse health outcomes. As part of an ongoing effort to identify molecular and physiologic triggers of inflammation in older adults, the investigators recently identified a highly significant inverse relationship between the anti-oxidant micronutrient selenium and the inflammatory mediator IL-6, as well as a significant relationship between selenium and all cause mortality in a population of community dwelling older women with selenium levels well below the mean for the overall American population. Based on our findings in older adults and on data from other studies that suggest that selenium interventions are effective in targeted populations with inflammatory conditions, the investigators hypothesize that selenium supplementation targeted to a population of older adults with increased inflammatory markers and low normal selenium levels will in the short term reduce inflammation as measured by serum IL-6, and in the long term will reduce the incidence and prevalence of inflammation associated poor health outcomes of frailty, disability, and mortality in vulnerable older adults.

ELIGIBILITY:
Inclusion Criteria:

* 70 years of age or older
* Able to provide written informed consent for screening and participation in the study

Exclusion Criteria:

* Taking a multi-vitamin containing 60 ug or more of Selenium more than once a week
* Have evidence of an active, untreated, acute inflammatory disease state such as rheumatoid arthritis, gout, or malignancy
* Taking any corticosteroids or the medications prednisone or methotrexate

Ages: 70 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 182 (Actual)
Dates: Start 2006-02 (Actual); Primary Completion 2012-01-20 (Actual); Study Completion 2012-01-20 (Actual)

PRIMARY OUTCOMES:
The effects of oral selenium supplementation on the inflammatory response in older adults with an increased IL-6 level and low normal selenium levels over an 8 week intervention period. | 8 weeks
  Serum Interleukin 6 (IL6)will be measured at baseline and every 2 weeks for the 8 weeks of the study using a standard, commercially available ELISA kit. Serum Selenium levels will also be measured at baseline and every 2 weeks for 8 weeks. The investigators hypothesize that as serum selenium levels increase with supplementation there will be a statistically significant decrease in serum IL6. IL6 levels should remain unchanged over 8 weeks in those taking the placebo.

SECONDARY OUTCOMES:
The effects of selenium supplementation on the activity of the selenium- dependent antioxidant enzyme glutathione peroxidase, and on altered protein production in older adults with increased serum IL-6 and low normal levels of selenium. | 8 weeks
  Glutathione peroxidase will be measured at baseline and at week 8. Glucose, Vitamin B-12, folate, methionine, and albumin will be measured in serum drawn at baseline and every 2 weeks for the 8 weeks of the study. the investigators hypothesize that levels of glutathione peroxidase and proteins may change significantly in participants taking selenium. There should be no significant changes in these parameters in those taking the placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy D Walston, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Walston J, Xue Q, Semba RD, Ferrucci L, Cappola AR, Ricks M, Guralnik J, Fried LP. Serum antioxidants, inflammation, and total mortality in older women. Am J Epidemiol. 2006 Jan 1;163(1):18-26. doi: 10.1093/aje/kwj007. Epub 2005 Nov 23. PMID 16306311
- [Background] Semba RD, Patel KV, Ferrucci L, Sun K, Roy CN, Guralnik JM, Fried LP. Serum antioxidants and inflammation predict red cell distribution width in older women: the Women's Health and Aging Study I. Clin Nutr. 2010 Oct;29(5):600-4. doi: 10.1016/j.clnu.2010.03.001. Epub 2010 Mar 23. PMID 20334961
- [Background] Ray AL, Semba RD, Walston J, Ferrucci L, Cappola AR, Ricks MO, Xue QL, Fried LP. Low serum selenium and total carotenoids predict mortality among older women living in the community: the women's health and aging studies. J Nutr. 2006 Jan;136(1):172-6. doi: 10.1093/jn/136.1.172. PMID 16365078